CLINICAL TRIAL: NCT00335504
Title: Randomized, Phase II Trial of Atorvastatin, RAFTILOSE Synergy 1, and Sulindac Among Patients at Increased Risk for Sporadic Colorectal Neoplasia
Brief Title: Atorvastatin Calcium, Oligofructose-Enriched Inulin, or Sulindac in Preventing Cancer in Patients at Increased Risk of Developing Colorectal Neoplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-00837; NCI-2009-00837 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000467755; MAY03-1-03 (Other: Mayo Clinic); MAY03-1-03 (Other: DCP); N01CN35000 (NIH); P30CA015083 (NIH)
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Results first posted 2013-02-08 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Colon Cancer; Precancerous Condition; Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Precancerous Conditions; Rectal Neoplasms | interventions — Sulindac; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Arm I (atorvastatin calcium) (Experimental): Patients receive oral atorvastatin once daily.
  Interventions: Drug: atorvastatin calcium; Other: laboratory biomarker analysis
- Arm II (sulindac) (Experimental): Patients receive oral sulindac twice daily.
  Interventions: Drug: sulindac; Other: laboratory biomarker analysis
- Arm III (oligofructose-enriched inulin) (Experimental): Patients receive oral oligofructose-enriched inulin (Raftilose Synergy 1) twice daily.
  Interventions: Drug: oligofructose-enriched inulin; Other: laboratory biomarker analysis
- Arm IV (placebo) (Placebo Comparator): Patients receive an oral placebo twice daily.
  Interventions: Drug: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: oligofructose-enriched inulin — Given orally
  Other Names: Beneo Synergy 1; Synergy 1
  Arms: Arm III (oligofructose-enriched inulin)
Drug: sulindac — Given orally
  Other Names: Aflodac; Algocetil; Clinoril; SULIN
  Arms: Arm II (sulindac)
Drug: placebo — Given orally
  Other Names: PLCB
  Arms: Arm IV (placebo)
Drug: atorvastatin calcium — Given orally
  Other Names: CI-981; Lipitor
  Arms: Arm I (atorvastatin calcium)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying atorvastatin calcium to see how well it works compared to oligofructose-enriched inulin, sulindac, or a placebo in preventing cancer in patients at increased risk of developing colorectal neoplasia. Chemoprevention is the use of certain drugs or substances to keep cancer from forming, growing, or coming back. The use of atorvastatin calcium, oligofructose-enriched inulin, or sulindac may stop cancer from forming in patients at increased risk of colorectal neoplasia. It is not yet known whether atorvastatin calcium, oligofructose-enriched inulin, or sulindac are more effective than a placebo in preventing cancer in patients at increased risk of developing colorectal neoplasia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Percent change in number of rectal aberrant cryptic foci (ACF) as measured by magnification chromoendoscopy

SECONDARY OBJECTIVES:

I. Screening for possible phase III testing II. Effects on proliferation (Ki67 expression) and apoptosis (caspase-3 expression) as measured by biopsy samples obtained from normal-appearing rectal mucosa at baseline and after completion of study treatment III. Correlation of endoscopic features with histologic characteristics of rectal ACF IV. Observation of the natural history of rectal ACF in patients receiving placebo V. Adverse events VI. Utilization of a biospecimen repository archive

OUTLINE: This is a multicenter, prospective, randomized, partially blinded, placebo-controlled study. Patients are stratified according to history of prior surgical resection of the colon (yes vs no) and number of rectal aberrant cryptic foci (ACF) (5-9 vs >= 10). Patients are randomized to 1 of 4 treatment arms.

ARM I: Patients receive oral atorvastatin calcium once daily.

ARM II: Patients receive oral sulindac twice daily.

ARM III (blinded arm): Patients receive oral oligofructose-enriched inulin (Raftilose Synergy 1) twice daily.

ARM IV (blinded arm): Patients receive an oral placebo twice daily.

In all arms, treatment continues for 6 months in the absence of unacceptable toxicity.

Tissue samples are collected at baseline and at the completion of study treatment. Tissue is examined by immunohistochemistry for proliferation (Ki67) and apoptosis (cleaved caspase-3).

After completion of study treatment, patients are followed at approximately 30 days.

ELIGIBILITY:
Criteria:

* ECOG performance status 0-2
* Platelet count >= 100,000/mm^3
* Fertile patients must agree to use effective contraception
* No history of inflammatory bowel disease (i.e., Crohn's disease or ulcerative colitis)
* No invasive malignancy within the past 5 years except nonmelanoma skin cancer or colorectal cancer
* No history of endoscopically-confirmed peptic ulcer disease
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to the study agents
* No history of chronic liver disease or unexplained persistent elevations of serum transaminases
* No history of allergic-type reactions, including asthma or urticaria, to aspirin or NSAIDs
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would preclude study compliance
* At least 6 weeks since prior oral corticosteroids
* Creatinine =< 1.5 times ULN
* Creatine phosphokinase =< 1.5 times ULN
* Not pregnant or nursing
* At least 6 weeks since prior statins
* At increased risk for developing sporadic colorectal neoplasia, as defined by 1 of the following:

  * History of colon cancer (excluding stage IV or Dukes' D tumors)
  * Must have completed prior adjuvant therapy for colon cancer >= 12 months ago
* History of colorectal adenomas, meeting any of the following criteria:

  * >= 1 cm in diameter
  * >= 3 in total number
  * Any component of villous morphology
  * High-grade dysplasia
* At least 5 rectal aberrant cryptic foci (ACF), by magnification chromoendoscopy, meeting both of the following criteria:

  * At least 5 aggregated crypts in a single grouping (maximum spacing between crypts must be =< 2 times the average crypt diameter)
  * Crypt diameter >= 1.5 times the diameter of surrounding normal crypts
* No history of rectal cancer, familial adenomatous polyposis, or hereditary nonpolyposis colorectal cancer
* Negative pregnancy test
* At least 6 months since prior and no concurrent regular use* of nonsteroidal anti-inflammatory drugs** (NSAIDs) or statins
* Concurrent aspirin at cardioprotective doses (=< 162.5 mg/day or 325 mg every other day) allowed
* No prior rectal surgery involving mucosal resection
* No prior pelvic radiation therapy
* No concurrent regular use* of cyclooxygenase-2 inhibitors
* No concurrent anticoagulant drugs (i.e., warfarin, heparin, clopidogrel bisulfate, or extended-release dipyridamole)
* No concurrent use of any of the following:

  * Fibrates (e.g., gemfibrozil or fenofibrate)
  * Cyclosporine
  * Erythromycin or macrolide antibiotics
  * Protease inhibitors
  * Azole antifungals
  * Diltiazem
  * Verapamil
  * Compounds containing niacin or nicotinic acid

    * Defined as 7 consecutive days for > 3 weeks OR > 21 days total during study participation
    * Patients may be eligible for study treatment after discontinuing NSAIDs for 12 weeks, at the discretion of their health care provider
* No other concurrent investigational agents
* No planned (or likely to require) clinically indicated colonoscopy or flexible sigmoidoscopy during study treatment
* Bilirubin =< 1.5 times ULN
* Hemoglobin >= lower limit of normal
* AST =< 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase =< 1.5 times ULN

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2006-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Limburg, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 142 subjects were pre-registered through 10 Cancer Prevention Network (CPN) member organizations from April 2006 to August 2008.
Pre-assignment Details: 57 subjects were excluded from the trial before assignment to groups: 13 did not have baseline Magnification chromoendoscopy (MCE), 33 had < 5 rectal ACF, 8 did not meet eligibility criteria, and 3 were withdrawn.
Groups:
- Arm I (Atorvastatin Calcium): Patients receive 20 mg tablet oral atorvastatin once daily.
- Arm II (Sulindac): Patients receive 150 mg tablet oral sulindac twice daily.
- Arm III (Oligofructose-enriched Inulin): Patients receive 6gm powder oral oligofructose-enriched inulin (Raftilose Synergy 1) twice daily.
- Arm IV (Placebo): Patients receive an oral placebo (maltodextrin powder) twice daily.
Period: Overall Study
Arm/Group | Arm I (Atorvastatin Calcium) | Arm II (Sulindac) | Arm III (Oligofructose-enriched Inulin) | Arm IV (Placebo)
Started | 22 | 21 | 20 | 22
Completed | 22 | 21 | 20 | 22
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Atorvastatin Calcium) | Arm II (Sulindac) | Arm III (Oligofructose-enriched Inulin) | Arm IV (Placebo) | Total
Number analyzed (Participants) | 22 | 21 | 20 | 22 | 85
Age, Continuous [Median (Full Range); unit: Years] | 61 [44 to 78] | 55 [41 to 74] | 64 [48 to 78] | 57 [44 to 72] | 58 [41 to 78]
Gender [Count of Participants; unit: Participants]
  Female | 5 | 9 | 8 | 7 | 29
  Male | 17 | 12 | 12 | 15 | 56
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 20 | 22 | 85
History of Surgical Resection [Number; unit: participants] — History of prior surgical resection of the colon: Yes vs. No
  participants
    Yes | 7 | 6 | 6 | 6 | 25
    No | 15 | 15 | 14 | 16 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Number of Rectal Aberrant Cryptic Foci (ACF) as Measured by Magnification Chromoendoscopy
Description: At the Pre-Intervention Evaluation, rectal ACF will be classified with respect to ACF number, crypt number, crypt size, tissue plane, staining intensity, and (optional) lumen shape for each subject. At the Post- Intervention Evaluation, these same parameters will be recorded and incident vs prevalent rectal ACF status will also be recorded. Compare each non-placebo arms versus the placebo arm to screen the three active study agents for possible phase III testing.
Time Frame: 6 months
Population: The population used for the analysis is patients having at least 5 rectal ACF and completing both the pre- and post-intervention MCE assessments and using intention to treat principles.
Measure: Mean (Standard Deviation); unit: percent change in number of ACF
Arm/Group | Arm I (Atorvastatin Calcium) | Arm II (Sulindac) | Arm III (Oligofructose-enriched Inulin) | Arm IV (Placebo)
Number analyzed (Participants) | 20 | 18 | 20 | 19
percent change in number of ACF | 8.4 (49.1) | -13.3 (55.4) | -8.8 (49.2) | -8.6 (48.8)
Statistical Analysis 1: Comparison: Arm I (Atorvastatin Calcium) vs Arm IV (Placebo); The study was designed to test the hypotheses of observing a 25% difference in % change ACF over baseline, between patients treated with atorvastatin compared to placebo. N=25 subjects per group yielded 93% power to detect this difference using a 2 sided t-test at significance level of 0.05. Non-parametric tests (eg, Wilcoxon Rank Sum) could be used if the statistical assumptions of the t-test were violated; Test type: Superiority or Other; p = 0.30, Wilcoxon (Mann-Whitney) — Adjusting for multiple comparisons yields 84% power to detect a difference of at least 25% in % change of ACF at the 0.016 level of significance and using a two-sample, 2-sided t-test
Statistical Analysis 2: Comparison: Arm II (Sulindac) vs Arm IV (Placebo); The study was designed to test the hypotheses of observing a 25% difference in % change ACF over baseline, between patients treated with sulindac compared to placebo. N=25 subjects per group yielded 93% power to detect this difference using a 2 sided t-test at significance level of 0.05. Non-parametric tests (eg, Wilcoxon Rank Sum) could be used if the statistical assumptions of the t-test were violated; Test type: Superiority or Other; p = 0.60, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Arm III (Oligofructose-enriched Inulin) vs Arm IV (Placebo); The study was designed to test the hypotheses of observing a 25% difference in % change ACF over baseline, between patients treated with oligofructose-enriched inulin compared to placebo. N=25 subjects per group yielded 93% power to detect this difference using a 2 sided t-test at significance level of 0.05. Non-parametric tests (eg, Wilcoxon Rank Sum) could be used if the statistical assumptions of the t-test were violated; Test type: Superiority or Other; p = 0.92, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Arm I (Atorvastatin Calcium); Signed Rank p-value for comparison of % change in ACF within each randomization arm; Test type: Superiority or Other; p = 0.59, Sign test
Statistical Analysis 5: Comparison: Arm II (Sulindac); Signed Rank p-value for comparison of % change in ACF within each randomization arm; Test type: Superiority or Other; p = 0.12, Sign test
Statistical Analysis 6: Comparison: Arm III (Oligofructose-enriched Inulin); Signed Rank p-value for comparison of % change in ACF within each randomization arm; Test type: Superiority or Other; p = 0.54, Sign test
Statistical Analysis 7: Comparison: Arm IV (Placebo); Signed Rank p-value for comparison of % change in ACF within each randomization arm; Test type: Superiority or Other; p = 0.41, Sign test

2. Secondary Outcome: Effects on Proliferation (Ki67 Expression).
Description: Tissue is examined by immunohistochemistry for Ki67. Measured by biopsy samples obtained from normal-appearing rectal mucosa at baseline and after completion of study treatment. Wilcoxon will be used to assess significant differences between the intervention arms.
Time Frame: Up to 6 months
Population: Patients with assay data from baseline and post-intervention biopsy samples of normal-appearing rectal mucosa.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Arm I (Atorvastatin Calcium) | Arm II (Sulindac) | Arm III (Oligofructose-enriched Inulin) | Arm IV (Placebo)
Number analyzed (Participants) | 16 | 17 | 13 | 15
Percent change | 6.5 (62.3) | 12.2 (52.8) | 34.7 (70.6) | 13.6 (44.1)
Statistical Analysis 1: Comparison: Arm I (Atorvastatin Calcium) vs Arm IV (Placebo); Wilcoxon Rank Sum p-value for comparison of % change in Ki67 between atorvastatin and placebo; Test type: Superiority or Other; p = 0.37, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm II (Sulindac) vs Arm IV (Placebo); Wilcoxon Rank Sum p-value for comparison of % change in Ki67 between sulindac and placebo; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm III (Oligofructose-enriched Inulin) vs Arm IV (Placebo); Wilcoxon Rank Sum p-value for comparison of % change in Ki67 between oligofructose-enriched inulin and placebo; Test type: Superiority or Other; p = 0.58, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Effects on Apoptosis (Caspase-3 Expression).
Description: Tissue is examined by immunohistochemistry for cleaved caspase-3. Measured by biopsy samples obtained from normal-appearing rectal mucosa at baseline and after completion of study treatment. Wilcoxon will be used to assess significant differences between the intervention arms.
Time Frame: Up to 6 months
Population: Patients with assay data from baseline and post-intervention biopsy samples of normal-appearing rectal mucosa.
Measure: Mean (Standard Deviation); unit: Percent change of caspase-3
Arm/Group | Arm I (Atorvastatin Calcium) | Arm II (Sulindac) | Arm III (Oligofructose-enriched Inulin) | Arm IV (Placebo)
Number analyzed (Participants) | 14 | 15 | 14 | 12
Percent change of caspase-3 | 106.0 (140.3) | 131.9 (154.1) | 120.5 (195.6) | 130.6 (81.8)
Statistical Analysis 1: Comparison: Arm I (Atorvastatin Calcium) vs Arm IV (Placebo); Wilcoxon Rank Sum p-value for comparison of % change in apoptosis between atorvastatin calcium and placebo; Test type: Superiority or Other; p = 0.26, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm II (Sulindac) vs Arm IV (Placebo); Wilcoxon Rank Sum p-value for comparison of % change in apoptosis between sulindac and placebo; Test type: Superiority or Other; p = 0.88, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm III (Oligofructose-enriched Inulin) vs Arm IV (Placebo); Wilcoxon Rank Sum p-value for comparison of % change in apoptosis between oligofructose-enriched inulin and placebo; Test type: Superiority or Other; p = 0.38, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Adverse Events.
Description: Defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with participation in a study, whether or not related to that participation. Graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 3.0. Number of adverse events per grade level.
Time Frame: Up to 30 days after completion of study treatment
Measure: Number; unit: adverse events
Arm/Group | Arm I (Atorvastatin Calcium) | Arm II (Sulindac) | Arm III (Oligofructose-enriched Inulin) | Arm IV (Placebo)
Number analyzed (Participants) | 22 | 21 | 20 | 22
adverse events
  Grade 1 | 11 | 12 | 10 | 15
  Grade 2 | 5 | 4 | 4 | 13
  Grade 3 | 2 | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: Start of treatment to 30 days past the end of treatment.
Description: Common Toxicity Criteria for Adverse Events (CTCAE) v3
Arm/Group | Arm I (Atorvastatin Calcium) | Arm II (Sulindac) | Arm III (Oligofructose-enriched Inulin) | Arm IV (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 15/22 | 14/21 | 12/20 | 19/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Atorvastatin Calcium) (N=22) | Arm II (Sulindac) (N=21) | Arm III (Oligofructose-enriched Inulin) (N=20) | Arm IV (Placebo) (N=22)
Constitutional Symptoms - Other Specify (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Auditory/Ear - Other Specify (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dermatology/Skin - Other Specify (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Endocrine - Other Specify (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (6) | 5 (6)
Gastrointestinal - Other Specify (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Heartburn (Gastrointestinal disorders) | 0 (0) | 4 (5) | 0 (0) | 3 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Infection - Other (Specify (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Headache (Nervous system disorders) | 2 (3) | 1 (3) | 2 (2) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (3) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary/Upper Respiratory - Other Specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Variation in endpoint measurement across sites, relatively small sample size, and rectal biomarker assessments only may have contributed to challenges in full data interpretation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less